CLINICAL TRIAL: NCT04275063
Title: Autism, Sport and Society: Conversations With Parents
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Midlands Psychology CIC (Other)
Responsible Party: Sponsor
Other Study IDs: MP/KA-2
Record Dates: First submitted 2020-02-17; First posted 2020-02-19 (Actual); Last update posted 2020-02-19 (Actual); Status verified 2020-02

CONDITIONS: Autism Spectrum Disorder
Keywords: ASC; Sport and physical activity; Parent perceptions
MeSH Terms: conditions — Autism Spectrum Disorder; Motor Activity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In order to examine the experience of children with ASC in physical activity at home, at school, and in the local community, parents of children with ASC will be asked a number of open ended interview questions. To see if these experiences are unique to parents of children ASC, parents of non-ASC children will also be interviewed to allow for these perspectives to be compared and contrasted.

DETAILED DESCRIPTION:
Background:

77% of boys and 80% of girls aged 5-15 in the UK fall below the national physical activity guidelines of 60 minutes of moderate to vigorous activity per day.

Research shows children with an Autism Spectrum Condition (ASC) are even less physically active than their neurotypical, age related peers and as a result are at increased risk of cardiovascular diseases, metabolic disorders, low self-esteem and depression. This physical activity gap has been shown to increase as children get older.

If a gap between the activity levels of children with ASC and the so called 'normal population' exists, there are a number of possible explanations for why this might be. Research points to either some facet of the autism spectrum causing difficulties engaging with a certain feature of a physical activity i.e. the physical environment in which activities take place which is difficult from the sensory point of view (noisy, busy, brightly lit) or lack of specific provision tailored towards children with ASC readily available in the local community. With repeated negative experiences, children and adults with ASC may come to believe these opportunities are 'not for them'.

To date, there has been limited research conducted on the attitudes of young people with ASC to sport and physical activity. The research that has been conducted has mainly focused on interviewing the young people themselves to gather their perspectives. However, little is known about their parent's perceptions of sports participation or if parents value being physically active themselves. This is of particular interest as parental modelling has been shown to be a predictor of children's PA behaviours with a positive correlation between adult and child PA levels. Furthermore, parents may offer additional insights into barriers of physical activity beyond that of their children and this information could help to advise the sports sector on how clubs and leisure centres could offer a better experience for children with ASC.

In order to examine the experience of children with ASC in physical activity at home, at school, and in the local community, parents of children with ASC will be asked a number of open ended interview questions. To see if these experiences are unique to parents of children ASC, parents of non-ASC children will also be interviewed to allow for these perspectives to be compared and contrasted.

ELIGIBILITY:
Inclusion Criteria:

* Parent of child with an Autism Spectrum Condition aged 5-15
* Parent of child aged 5-15

Exclusion Criteria:

* Parents with children with autism older than 15 or younger than 5
* Parents of children older than 15 or younger than 5

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: The sample will consist of 15 parents/carers of children with an ASC between the ages of 5-15 and 15 parents/carers of children without ASC between the ages of 5-15.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2020-03-01 (Estimated); Primary Completion 2020-08-01 (Estimated); Study Completion 2020-08-01 (Estimated)

PRIMARY OUTCOMES:
Child Physical Activity and Parent Attitudes to Sport: Parent Questionnaire | 1 year
  Qualitative interview for parents of children with and without autism spectrum disorders to examine perceptions of their chid's physical activity at school, at home and in the local community. To be conducted on one occasion.
  The interview guide is grouped into 4 sections: current activity levels, parent perceptions on activity and their local community, physical activity in school, and opinions on the sports sector and how it can be changed.
  Examples of questions include "What types of physical activity does your child take part in currently?" and "What has been your child's experiences of P.E in school?"

CONTACTS AND LOCATIONS:
Overall Officials: James Smolinski, MSc, Principal Investigator — Midlands Psychology CIC

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cridland EK, Jones SC, Magee CA, Caputi P. Family-focused autism spectrum disorder research: a review of the utility of family systems approaches. Autism. 2014 Apr;18(3):213-22. doi: 10.1177/1362361312472261. Epub 2013 Oct 3. PMID 24092840
- [Background] Healy, S., Msetfi, R., & Gallagher, S. (2013). 'Happy and a bit nervous': The experiences of children with autism in physical education. British Journal of Learning Disabilities, 41(3), 222-228.
- [Background] Kohl HW 3rd, Hobbs KE. Development of physical activity behaviors among children and adolescents. Pediatrics. 1998 Mar;101(3 Pt 2):549-54. PMID 12224661
- [Background] Memari, A. H., Kordi, R., Ziaee, V. et al. (2012). Weight status in Iranian children with autism spectrum disorders: Investigation of underweight, overweight and obesity. Research in Autism Spectrum Disorders, 6(1), 234-239.
- [Background] Padgett, D. K. (1998). Qualitative methods in social work research: Challenges and rewards. Thousand Oaks, CA: Sage.
- [Background] Pan CY. Objectively measured physical activity between children with autism spectrum disorders and children without disabilities during inclusive recess settings in Taiwan. J Autism Dev Disord. 2008 Aug;38(7):1292-301. doi: 10.1007/s10803-007-0518-6. Epub 2007 Dec 18. PMID 18157623
- [Background] Public Health England (2016). Health matters: getting every adult active every day. [online] Available at: https://www.gov.uk/government/publications/health-matters-getting-every-adult-active-every-day/health-matters-getting-every-adult-active-every-day [Accessed 20 Aug. 2019].
- [Background] Rimmer JH, Yamaki K, Lowry BM, Wang E, Vogel LC. Obesity and obesity-related secondary conditions in adolescents with intellectual/developmental disabilities. J Intellect Disabil Res. 2010 Sep;54(9):787-94. doi: 10.1111/j.1365-2788.2010.01305.x. Epub 2010 Jul 12. PMID 20630017